CLINICAL TRIAL: NCT06369636
Title: Comparison of El-Ganzouri Risk Index and Airway Ultrasonographic Evaluation In Terms of Predicting Difficult Intubation in Patients Undergoing Thyroid Surgery
Brief Title: Comparison of El-Ganzouri Risk Index and Airway Ultrasonographic Evaluation in Thyroid Surgery
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: myucesu
Record Dates: First submitted 2024-04-04; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Surgery; Difficult Intubation
Keywords: Thyroid Surgery; El-Ganzouri Risk Index; Airway Ultrasonography; Difficult Intubation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Difficult Intubation Expected: Patients whose EGRI scores are equal or greater than 4, or whose skin to epiglottis measurement are greater than 18 mm, skin to hyoid bone measurement are greater than 14 mm, skin to anterior commissure of vocal cords are greater than 13 mm, tongue thickness are greater than 60 mm and tongue volume greater than 100 cm3.
  Interventions: Procedure: Thyroid Surgery
- Difficult Intubation Not Expected: Patients who do not meet the criteria just mentioned
  Interventions: Procedure: Thyroid Surgery

INTERVENTIONS:
Procedure: Thyroid Surgery — EGRI scores and airway ultrasonographic values will be recorded in patients who undergo thyroid surgery.

SUMMARY:
The primary purpose of this prospective observational study was to compare these tests used to predict difficult intubation in patients undergoing thyroid surgery. Secondarily; By comparing these tests, we aim to find the test that best predicts difficult intubation and to determine the incidence of difficult intubation in patients who will undergo thyroid surgery.

DETAILED DESCRIPTION:
Patients' demographic information (age, gender, American Society of Anesthesiologists (ASA) classification, STOP-BANG score(snoring, feeling tired, observed apnea, hypertension, obesity, age, neck circumference and gender), body mass index) and thyroid ultrasonographic measurement will be recorded.

At the preoperative visit, patients will be evaluated for El-Ganzouri Risk Index (EGRI) scores (mouth opening, thyromental distance, mallampati score, neck movement limitation, presence of prognathia, body weight and history of difficult intubation) and for airway ultrasonography (skin-epiglottis distance, skin-hyoid bone distance, skin-vocal cord distance, tongue thickness and tongue volume values).

After this information is recorded, patients will be grouped as those expected difficult intubation and those who are not. After the patients are taken to the operating table and monitored, vascular access will be opened, standard anesthesia induction will be applied to the patients by the room specialist, and laryngoscopy and endotracheal intubation will be performed by the trained (>2 years experienced) anesthesiologist. If Intubation Difficulty Scale (IDS) score will be greater than 5, patient will be considered difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA scores 1-3
* Patients between 18-65 age
* Patients who undergo thyroid surgery

Exclusion Criteria:

* Patients who do not accept to participate the research
* Patients under age 18 and over age 65
* Pregnant patients
* Patients who undergo surgery due to emergency medical conditions (such as hematoma, thyroid crisis or myxedema coma)
* Patients with airway malformations
* Patients with a high risk of aspiration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 120 patients, with ASA scores 1-3, aged between 18-65 years who undergo thyroid surgery will be included.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Compare EGRI and airway ultrasonographic parameters | Up to 6 months, until the end of the study
  Compare EGRI and airway ultrasonography for predicting difficult intubation in patients who undergoing thyroid surgery

SECONDARY OUTCOMES:
Find which is the best test predicts difficult intubation | Up to 6 months, until the end of the study
  by comparing these tests to decide which test is the best predictor for difficult intubation in thyroid surgery
Finding the incidence of difficult intubation in thyroid surgery | Up to 6 months, until the end of the study
  Determine the incidence of difficult intubation in thyroid surgery

CONTACTS AND LOCATIONS:
Overall Officials: Şeref Çelik, Principal Investigator — Ankara Bilkent City Hospital, Algology Clinic
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Langenstein H, Cunitz G. [Difficult intubation in adults]. Anaesthesist. 1996 Apr;45(4):372-83. doi: 10.1007/s001010050274. German. PMID 8702056
- [Result] Bacuzzi A, Dionigi G, Del Bosco A, Cantone G, Sansone T, Di Losa E, Cuffari S. Anaesthesia for thyroid surgery: perioperative management. Int J Surg. 2008;6 Suppl 1:S82-5. doi: 10.1016/j.ijsu.2008.12.013. Epub 2008 Dec 13. PMID 19195946
- [Result] Adhikari S, Zeger W, Schmier C, Crum T, Craven A, Frrokaj I, Pang H, Shostrom V. Pilot study to determine the utility of point-of-care ultrasound in the assessment of difficult laryngoscopy. Acad Emerg Med. 2011 Jul;18(7):754-8. doi: 10.1111/j.1553-2712.2011.01099.x. Epub 2011 Jun 27. PMID 21707828
- [Result] Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, Fiadjoe JE, Greif R, Klock PA, Mercier D, Myatra SN, O'Sullivan EP, Rosenblatt WH, Sorbello M, Tung A. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022 Jan 1;136(1):31-81. doi: 10.1097/ALN.0000000000004002. PMID 34762729
- [Result] Zheng Z, Ma W, Du R. Effectiveness and validity of midsagittal tongue cross-sectional area and width measured by ultrasound to predict difficult airways. Minerva Anestesiol. 2021 Apr;87(4):403-413. doi: 10.23736/S0375-9393.20.14769-2. Epub 2021 Feb 16. PMID 33591134